CLINICAL TRIAL: NCT03165955
Title: A Clinical Study to Determine the Pharmacokinetics of Oraxol in Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Health Hope Pharma (Industry)
Collaborators: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-007; U1111-1176-4228 (Other: ICTRP)
Record Dates: First submitted 2017-05-14; First posted 2017-05-24 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Breastcancer
Keywords: breast cancer; paclitaxel
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Oraxol (Experimental): Subjects will receive Oraxol 205 mg/m2 daily x 3 days weekly for up to 16 weeks.
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — HM30181 methanesulfonate monohydrate - supplied as 15-mg HM30181AK-US tablets, Paclitaxel - supplied as 30-mg capsules
  Other Names: HM30181 methanesulfonate monohydrate; Oral paclitaxel capsules

SUMMARY:
This is a multicenter, open-label, single-arm PK study in patients for whom paclitaxel treatment is indicated.

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm PK study in approximately 24 breast cancer patients for whom paclitaxel treatment is indicated. The study contains 3 periods: the Screening / Baseline Period, the Treatment Period, and the Follow-up Period. A Final Visit will occur within 7 days of the last dose of study treatment. If subjects achieve stable disease (SD), partial response (PR), or complete response (CR) at the end of the Treatment Period, they may continue Oraxol treatment in a separate extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Women ≥18 years of age on day of consent
3. Breast cancer in patients for whom treatment with IV paclitaxel at 80 mg/m2 as monotherapy has been recommended by their oncologist
4. Measurable disease as per RECIST v1.1 criteria
5. Adequate hematological status as demonstrated by not requiring transfusion support or granulocyte-colony stimulating factor (G-CSF) maintain:

   * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
   * Platelet count ≥100 x 10^9/L
   * Hemoglobin (Hgb) ≥9 g/dL
6. Adequate liver function

   * Total bilirubin of ≤1.5 mg/dL
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if liver metastasis is present
   * Alkaline phosphatase (ALP) ≤3 x ULN or ≤5 x ULN if bone metastasis is present
   * Gamma glutamyl transferase (GGT) <10 x ULN
7. Adequate renal function as demonstrated by serum creatinine ≤1.5 x ULN
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
9. Life expectancy of at least 3 months
10. Willing to fast for 6 hours before and 2 hours after Oraxol administration on all treatment days
11. Willing to abstain from alcohol consumption for 3 days before the first dose of study drug through the completion of the second inpatient PK sampling period
12. Willing to refrain from caffeine consumption for 12 hours before each inpatient dosing period through the completion of protocol-specified PK sampling for that week
13. Subjects must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for 30 days after their last dose of assigned study treatment.
14. Subjects who are of childbearing potential must have a negative serum pregnancy test at Screening and within 96 hours before dosing.

Exclusion Criteria:

1. Have not recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous investigational products (IPs)
2. If previously treated with a taxane (paclitaxel or docetaxel) as part of anthracycline-based adjuvant chemotherapy or for metastatic disease, the subject relapsed less than 1 year following treatment
3. Subjects unable to swallow study medication in its intact form or have clinically significant malabsorption syndrome
4. Only site of metastatic disease is unmeasurable according to RECIST v1.1 criteria
5. Known CNS metastasis, including leptomeningeal involvement
6. Received IPs within 14 days or 5 half-lives of the first study dosing day, whichever is longer
7. Are currently receiving other medications intended for the treatment of their malignancy
8. Women who are pregnant or breastfeeding
9. Taking prohibited medications:
10. Use of warfarin. Subjects receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or any concomitant illness or social situation that would limit compliance with study requirements
12. Known allergic reaction or intolerance to study medication components
13. Known allergic reaction or intolerance to contrast media
14. Subjects who, in the Investigator's opinion, are not suitable for participation in this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsu-Yi Chao, MD, DMS, PhD, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (6):
- Taiwan (6):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans Generla Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Shuang Ho Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dai MS, Chao TC, Chiu CF, Lu YS, Shiah HS, Jackson CGCA, Hung N, Zhi J, Cutler DL, Kwan R, Kramer D, Chan WK, Qin A, Tseng KC, Hung CT, Chao TY. Oral paclitaxel and encequidar in patients with breast cancer: a pharmacokinetic, safety, and antitumor activity study. Ther Adv Med Oncol. 2023 Jul 21;15:17588359231183680. doi: 10.1177/17588359231183680. eCollection 2023. PMID 37492633

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 31 subjects were screened; 3 subjects were screen failures and were not included in the analysis
Groups:
- Oraxol (Oral Paclitaxel Plus HM30181): Oraxol 205 mg/m2 daily x 3 days weekly for up to 16 weeks.
Period: Screening/Baseline
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Started | 31
Completed | 28
Not Completed | 3
Period: Treatment
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Started | 28
Completed | 20
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Progressive disease | 3

BASELINE CHARACTERISTICS:
Population: A total of 31 subjects were screened; 3 subjects were screen failures and were not included in the analysis
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 28
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 28
ECOG [Count of Participants; unit: Participants]
  0 | 24
  1 | 4

OUTCOME MEASURES:

1. Primary Outcome: PK Parameters for paclitaxel_AUC (0-52)
Description: PK parameters were summarized using the mean, SD
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
ng*hr/mL
  Week 1 | 3419 (1475)
  Week 4 | 3224 (1150)

2. Primary Outcome: PK Parameters for paclitaxel_Cmax
Description: PK parameters were summarized using the mean, SD
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
ng/mL
  Week 1 | 366 (143)
  Week 4 | 356 (140)

3. Primary Outcome: PK Parameters for paclitaxel_Ctrough(24)
Description: PK parameters were summarized using the mean, SD
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
ng/mL
  Week 1 | 11.0 (4.0)
  Week 4 | 12.5 (8.7)

4. Primary Outcome: PK Parameters for paclitaxel_Ctrough(48)
Description: PK parameters were summarized using the mean, SD
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
ng/mL
  Week 1 | 12.6 (4.3)
  Week 4 | 11.7 (3.3)

5. Primary Outcome: PK Parameters for paclitaxel_Cmax(0-24)
Description: PK parameters were summarized using the mean, SD
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
ng/mL
  Week 1 | 312 (132)
  Week 4 | 267 (135)

6. Primary Outcome: PK Parameters for paclitaxel_Cmax(24-48)
Description: PK parameters were summarized using the mean, SD
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
ng/mL
  Week 1 | 274 (144)
  Week 4 | 298 (127)

7. Primary Outcome: PK Parameters for paclitaxel_Cmax(48-52)
Description: PK parameters were summarized using the mean, SD
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
ng/mL
  Week 1 | 287 (144)
  Week 4 | 288 (144)

8. Primary Outcome: PK Parameters for paclitaxel_tmax(0-24)
Description: PK parameters were summarized using the median, minimum, maximum
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Median (Full Range); unit: hour
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
hour
  Week 1 | 1.05 [0.97 to 2.12]
  Week 4 | 1.07 [0.93 to 2.12]

9. Primary Outcome: PK Parameters for paclitaxel_tmax(24-48)
Description: PK parameters were summarized using the median, minimum, maximum
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Median (Full Range); unit: hour
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
hour
  Week 1 | 25.03 [24.47 to 27.03]
  Week 4 | 25.00 [22.78 to 27.33]

10. Primary Outcome: PK Parameters for paclitaxel_tmax(48-52)
Description: PK parameters were summarized using the median, minimum, maximum
Time Frame: PK sampling timepoints: predose, and at 1, 2, 3, and 4 hours after dosing of Day 1, 2, 3 at Week 1 and 4
Population: Twenty-five subjects completed 2-period PK assessment.
Measure: Median (Full Range); unit: hour
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 25
hour
  Week 1 | 49.02 [48.22 to 51.03]
  Week 4 | 49.03 [47.05 to 51.05]

11. Secondary Outcome: Safety of Oraxol in Breast Cancer Patients
Description: Safety was assessed by evaluating treatment-emergent adverse events (TEAEs) including SAEs, laboratory evaluations (hematology, blood chemistry, and urinalysis), vital signs, physical examinations, and electrocardiograms (ECGs).
Time Frame: From enrollment through study completion, approximately 17 weeks
Population: Safety Analysis Population included all subjects who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 28
Participants
  Subjects with At Least One TEAE | 27
  TEAE leading to dose interruption or reduction | 19
  TEAE leading to study drug discontinuation | 2
  TEAE leading to discontinuation from the study | 2
  Serious TEAE | 8
  TEAE related to Oraxol | 27
  TEAE related to progression of disease | 4
  Death | 1
  TEAE with action taken for other treatments | 24
  Subjects with At Least One Grade ≥3 TEAE | 19

12. Secondary Outcome: Response Rate
Description: Tumor response rate and 95% confidence interval (CI) were evaluated based on the number of subjects with any post-baseline CR or PR per RECIST 1.1 as assessed by the Investigator and the ICRRC.
Time Frame: From baseline through study completion, around 21 weeks
Population: The Response Evaluable Population included all subjects who received at least 1 dose of study treatment and had at least 1 post treatment tumor response evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 26
Participants
  Investigator Assessment: Complete response (CR) | 0
  Investigator Assessment: Partial response (PR) | 11
  Investigator Assessment: Stable disease (SD) | 13
  Investigator Assessment: Progressive disease (PD) | 1
  Investigator Assessment: Non-evaluable (NE) | 1
  ICRRC Assessment: number analyzed (Participants) | 25
  ICRRC Assessment: Complete response (CR) | 0
  ICRRC Assessment: Partial response (PR) | 10
  ICRRC Assessment: Stable disease (SD) | 12
  ICRRC Assessment: Progressive disease (PD) | 3
  ICRRC Assessment: Non-evaluable (NE) | 0

13. Secondary Outcome: Progression-free Survival
Description: PFS was analyzed based on the Response Evaluable Population. The Kaplan-Meier (KM) method was used to estimate the medians of these variables with 95% CIs.
  The Response Evaluable Population included all subjects who received at least 1 dose of study treatment and had at least 1 posttreatment tumor response evaluation
Time Frame: From baseline through study completion, around 21 weeks
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 26
weeks
  Investigator Assessment | NA [NA to NA] — NA indicates that it cannot be estimated based on the data. Median OS is not reached
  ICRRC Assessment: number analyzed (Participants) | 25
  ICRRC Assessment | 15.86 [15.00 to NA] — NA indicates that it cannot be estimated based on the data. Median OS is not reached

14. Secondary Outcome: Overall Survival
Description: OS was analyzed based on the Response Evaluable Population. The Kaplan-Meier (KM) method was used to estimate the medians of these variables with 95% CIs.
  The Response Evaluable Population included all subjects who received at least 1 dose of study treatment and had at least 1 posttreatment tumor response evaluation
Time Frame: From baseline through study completion, around 21 weeks
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
Number analyzed (Participants) | 26
weeks | NA [NA to NA] — NA indicates that it cannot be estimated based on the data. Median OS is not reached

ADVERSE EVENTS:
Time Frame: An AE was any untoward medical occurrence in a subject or clinical investigation subject, and included events occurring from the time a subject signed the ICF through the last subject contact. The period is up to 21 weeks.
Arm/Group | Oraxol (Oral Paclitaxel Plus HM30181)
All-Cause Mortality (participants affected / at risk) | 1/28
Serious Adverse Events (participants affected / at risk) | 8/28
Other Adverse Events (participants affected / at risk) | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oraxol (Oral Paclitaxel Plus HM30181) (N=28)
Neutropenia (Blood and lymphatic system disorders) | 3 (8)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (2)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oraxol (Oral Paclitaxel Plus HM30181) (N=28)
Diarrhoea (Gastrointestinal disorders) | 16 (28)
Nausea (Gastrointestinal disorders) | 9 (20)
Vomiting (Gastrointestinal disorders) | 4 (5)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Mouth ulceration (Gastrointestinal disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 16 (62)
Anaemia (Blood and lymphatic system disorders) | 6 (16)
Leukopenia (Blood and lymphatic system disorders) | 3 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 5 (13)
Aspartate aminotransferase increased (Investigations) | 5 (12)
Blood lactate dehydrogenase increased (Investigations) | 2 (8)
White blood cell count decreased (Investigations) | 2 (5)
Neuropathy peripheral (Nervous system disorders) | 4 (9)
Dizziness (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 2 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (3)
Urinary tract infection (Infections and infestations) | 2 (2)
Fatigue (General disorders) | 2 (3)
Malaise (General disorders) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3)
Insomnia (Psychiatric disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT03165955/Prot_SAP_003.pdf